CLINICAL TRIAL: NCT06949826
Title: A Single-institution, Parallel, Double-blinded, Randomized Study Assessing the Safety and Efficacy of Transdermal Buprenorphine as a Post-operative Analgesic in Opioid-Naive Patients After Ankle Fracture Surgery
Brief Title: Buprenorphine as a Post-operative Analgesic in Opioid-Naive Patients After Ankle Fracture Surgery
Acronym: BAFA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jenna-Leigh Wilson (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other); Washington University Institute of Clinical and Translational Sciences (Unknown)
Responsible Party: Sponsor-Investigator, Jenna-Leigh Wilson, Assistant Professor of Orthopaedic Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202406162
Record Dates: First submitted 2025-04-11; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative; Ankle Fracture Surgery; Opioid Use Disorder; Opioid Dependence; Opioid Analgesia
Keywords: Buprenorphine; Postoperative pain; Transdermal buprenorphine; Ankle fracture surgery; Ankle fracture; Opioid-naive patient; ORIF Ankle Fracture; Opioid use disorder; Opioid Addiction; Buprenorphine for postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders; Ankle Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buprenorphine Transdermal System (Experimental): Participants in this arm will be treated with the transdermal buprenorphine system (a transdermal patch) that is applied in the pre-operative holding area. Aside from being treated with the transdermal buprenorphine system, their care will otherwise be in accordance with the standard of care following ankle fracture surgery.
  Interventions: Drug: Buprenorphine Transdermal System
- Placebo Patch (Placebo Comparator): Participants in this arm will be treated with a placebo patch that is applied in the pre-operative holding area. Aside from the placebo patch, their care will otherwise be in accordance with the standard of care following ankle fracture surgery.
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: Buprenorphine Transdermal System — The buprenorphine transdermal system is unique from other interventions in the study, as it is the experimental drug in the study. The buprenorphine transdermal system will be applied in the pre-operative holding area. Aside from the buprenorphine transdermal system, participants assigned to this intervention will otherwise receive the standard of care in their post-operative pain management following ankle fracture surgery.
  Arms: Buprenorphine Transdermal System
Drug: Placebo Patch — The placebo patch is unique from other interventions in the study, as it is the placebo drug in the study. The placebo patch will be applied in the pre-operative holding area. Aside from the placebo patch, participants assigned to this intervention will otherwise receive the standard of care in their post-operative pain management following ankle fracture surgery.
  Arms: Placebo Patch

SUMMARY:
Addictive full-agonist opioids, like oxycodone and hydrocodone, are often used to treat pain after surgery. However, these full-agonist opioids can be very addictive. After ankle fracture surgery, about 1 in 5 patients that did not take opioids before surgery become addicted to opioids after surgery. Buprenorphine is an opioid with unique properties that may offer a way to reduce the number of patients that become addicted to opioids after surgery. Buprenorphine has good analgesic (painkilling) effects. It is also thought to be less addictive and cause less of a high than full-agonist opioids, like oxycodone and hydrocodone. This project's goal is to determine if transdermal buprenorphine can safely and effectively control pain after ankle fracture surgery. This study will be a pilot study, which sets the stage for future studies that investigate whether buprenorphine can reduce the rate that patients become addicted to opioids after surgery. This study's multidisciplinary team will divide patients into two groups. Participants in one group will be treated with a 7-day transdermal buprenorphine patch (where the buprenorphine is slowly absorbed through the skin over 7 days). Participants in the other group will be treated with a placebo patch. A placebo has no drug in it, it just looks like the buprenorphine patch. Aside from the buprenorphine patch or placebo patch, both groups' pain management plans will be the same as if they were not in the study. Over the first week after surgery, the investigators will measure the amount of full-agonist opioids (for example, oxycodone or hydrocodone) that participants consume, participants' pain scores, the frequency of side effects related to opioids, and the number of calls and patient portal messages to the clinic for uncontrolled pain. The investigators will also assess whether participants are continuing to use opioids 3 months after surgery for pain related to their ankle fracture.

DETAILED DESCRIPTION:
Addictive full-agonist opioids, like oxycodone, remain a staple of post-operative analgesia after many types of surgery. However, perioperative exposure to opioid analgesics risks addiction in up to 7% of cases. Moreover, opioid overdoses kill over 80,000 in the United States (US) annually. Buprenorphine, a partial-agonist of the μ-opioid receptor and an antagonist of the κ-opioid receptor, may be able to safely function as a post-operative analgesic, reducing our reliance on full-agonist opioids post-operatively. Compared to full-agonist opioids, buprenorphine has a favorable safety profile. It has been hypothesized that buprenorphine's unique pharmacodynamics give it a lower addictive potential compared to full-agonist opioids. Moreover, it endows a ceiling on respiratory depression, has reduced dysphoric and psychotomimetic effects, and does not result in immunosuppression at therapeutic analgesic doses. International studies have suggested that transdermal buprenorphine is noninferior to tramadol, transdermal fentanyl, and oral celecoxib in the management of acute post-operative pain in opioid-naïve patients following orthopaedic surgery. However, the efficacy of buprenorphine for postoperative analgesia has never been studied in the United States, whose population has different beliefs and expectations surrounding pain control when compared to international populations. The major goal of this project is to determine the safety and efficacy of transdermal buprenorphine for postoperative analgesia, as a first step toward exploring the ability of buprenorphine to mitigate the incidence of opioid dependence in the postoperative setting.

This study will assess whether buprenorphine can reduce the use of full-agonist opioids following ankle fracture surgery. Approximately one in five opioid-naïve patients undergoing ankle fracture surgery continue to use opioids 3 to 6 months out from surgery, suggesting that this population is relatively susceptible to developing post-operative opioid dependence. The investigators will divide patients into two groups. One group will be treated with a 7-day transdermal buprenorphine patch. The other will be treated with a placebo patch. Both groups will otherwise receive a post-operative pain management regimen that is in accordance with the standard of care. The investigators hypothesize that participants treated with the buprenorphine patch will experience improved analgesia with the use fewer full-agonist opioids following ankle fracture surgery than those treated with the placebo patch. This hypothesis will be tested with the following aims.

Specific Aim 1: To measure the analgesic effect of buprenorphine on post-operative analgesia. In this Aim, the investigators will test the hypothesis that use of buprenorphine patches will reduce the average pain scores and consumption of full-agonist opioids after ankle fracture surgery. In sub-Aim 1.1, the investigators will quantify postoperative pain by monitoring participants' visual analog scale pain scores and full-agonist opioid consumption over the first post-operative week. In sub-Aim 1.2, the investigators will track the number of episodes of breakthrough pain in the hospital, the number of calls to the clinic with a chief complaint of uncontrolled pain, and the number of presentations to an emergency department for uncontrolled surgery-related pain.

Specific Aim 2: To examine the safety of buprenorphine as a post-operative analgesic following ankle fracture surgery. In this Aim, the investigators will test the hypothesis that participants treated with buprenorphine patches will experience fewer adverse events related to opioid exposure compared to those treated with placebo patches. The investigators will monitor for adverse effects of buprenorphine and full-agonist opioids, including respiratory depression, constipation, nausea, and vomiting. The investigators will track the number of presentations to an emergency department with a diagnosis of opioid toxicity. For pilot data, the investigators will also monitor use of opioids for analgesia at the 3-month postoperative time point as a secondary outcome.

This study assesses whether buprenorphine safely reduces full-agonist opioid use after orthopaedic surgery. Completion of the Aims of this study will permit future studies assessing whether buprenorphine comprises a less-addictive alternative for postoperative analgesia compared to full-agonist opioids. Annually, there are 40-50 million major surgeries performed in the US. As 6-7% of opioid-naïve patients develop long-term opioid use after major surgery, exploring avenues to decrease the impact of post-operative analgesia on the opioid epidemic is critical.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patient is 18 years of age or older
* Patient is undergoing single stage ORIF of an ankle fracture
* Patient is English-speaking

EXCLUSION CRITERIA:

* Patient is under 18 years of age
* Patient's ankle fracture is treated with external fixation
* Patient has a concomitant osseous or visceral injury
* Patient has a history of opioid use disorder or a current diagnosis of opioid use disorder
* Patient has a history of alcohol use disorder or a current diagnosis of alcohol use disorder
* Patient was taking opioid medication or narcotic drugs prior to their injury
* Patient has a current active malignancy
* Patient is taking a medication that carries a prohibitively high risk of drug-drug interaction with buprenorphine, hydrocodone, or oxycodone in the view of their treating physician or nurse anesthetist
* Patient has an anaphylactic allergy to buprenorphine, hydrocodone, or oxycodone
* Patient is not English-speaking
* Patient is pregnant
* Patient is unable to complete pain diary or communicate pain scores
* Patient is incarcerated
* Patient has a Gustilo-Anderson Type III open fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Pain Scores | Postoperative days 1-8, 21, 90.
  After surgery, visual analog pain scores with movement and at rest will be reported by the patient in a pain diary. In admitted patients, visual analog pain scores will be recorded by the bedside nurse. Visual analog pain scores are rated from 0-10. A score of 0 represents that the patient has no pain. A score of 10 represents excruciating pain.
Morphine Milligram Equivalents of Full-agonist Opioid Consumed | Post-operative days 0-7. First post-operative clinic visit (approximately 3 weeks after surgery).
  After surgery, patients will record the total amount of opioid medication they consumed during the first post-operative week in their pain diary. In admitted patients, the electronic medical record will be reviewed to determine the morphine milligram equivalents of opioid consumed while admitted. Patients will also bring all their bottles and opioid prescriptions to their first post-operative clinic visit, at which point their total opioid consumption between surgery and their first post-operative clinic visit will be recorded by the researchers.
Hospital Readmissions due to Opioid Toxicity | From patch application to post-operative day 21
  The researchers will track the number of hospital readmissions secondary to opioid toxicity.
Emergency Department Presentations due to Opioid Toxicity | From patch application to post-operative day 21
  The researchers will track the number of presentations to the emergency department with a chief complaint of opioid toxicity.
Emergency Department Presentations due to Uncontrolled Pain | From patch application through post-operative day 21.
  The investigators will track the number of emergency department presentations, with a chief complaint of uncontrolled post-operative pain.
Hospital Readmissions due to Uncontrolled Post-operative Pain | From patch application through post-operative day 21.
  The investigators will track the number of hospital readmissions due to uncontrolled post-operative pain.
Adverse Effects Related to Opioid Medication | Post-operative days 1-8, 21.
  After surgery, patients will record whether they have symptoms of constipation, nausea, vomiting, drowsiness, or anything other symptoms potentially related to their opioid medication. The frequency and types of adverse effects will be recorded by the study researchers.

SECONDARY OUTCOMES:
Morphine Milligram Equivalents of Full-Agonist Opioids Administered in Perioperative Setting | Perioperative/Periprocedural
  Review of the medication administration record will be performed to calculate the morphine milligram equivalents of opioid medication administered during ankle fracture surgery and in the post-operative recovery unit.
Time from Surgery Completion to Discharge | Perioperative/periprocedural
  For patients undergoing outpatient surgery, review of the electronic medical record will be performed to determine the time from surgery completion to discharge.
Hospital Length of Stay | From the completion of ankle fracture surgery to hospital discharge.
  For patients being admitted to the hospital to recover after ankle fracture surgery, review of the electronic medical record will be performed to determine the average hospital length of stay for each group.
Number of Breakthrough Pain Episodes while Inpatient | Post-operative day 0 through hospital discharge
  For patients admitted after surgery, the number of breakthrough pain episodes while inpatient will be determined. A breakthrough pain episode will be defined as a sudden, severe, brief pain occurring in the setting go f adequately controlled mild-moderate background pain. It will be denoted by the administration of a medication in the inpatient setting with an indication of "for breakthrough pain."
Quality of Recovery after Anesthesia 15-Question Survey | Post-operative day 7
  Patients will complete the quality of recovery after anesthesia 15-question survey. Scores range from 0 to 150. A score of 0 represents a poor recovery after anesthesia. A score of 150 represents an excellent recover after anesthesia.
Telephone Calls and MyChart Messages to Clinic or Call Center with a Chief Complaint of Uncontrolled Pain | Post-operative days 0-21.
  Review of the electronic medical record will be performed to record the average number of telephone calls and MyChart messages to the orthopaedic surgery clinic or call center with a chief complaint of uncontrolled pain.
Opioid Medication Prescriptions - Number and Total Morphine Milligram Equivalents Prescribed | From the time of injury through post-operative day 90.
  The researchers will review the electronic medical record to record the number of opioid medication prescriptions requested and filled by the patient.
Drug Liking and Economic Choice Survey | Post-operative days 7, 21, 90
  Patients will be asked by questionnaire how much they liked their buprenorphine vs placebo patch and oral narcotic prescriptions, as well as how much they would pay for their buprenorphine vs placebo patch and oral full-agonist opioid prescription.
Patient Satisfaction with Post-operative Pain Control | Post-operative days 7, 21
  Patient satisfaction with their post-operative pain control will be recorded by questionnaire in the form of a Likert scale.
Rate of Persistent Opioid Use | Post-operative day 90
  Approximately three months after surgery, patients will record whether they are continuing to take opioids/narcotics for pain related to their ankle fracture surgery.
Prescription Pain Medication Misuse Short Form 7a Scores | Post-operative day 90
  Patients will complete the PROMIS Prescription Pain Medication Misuse Short Form 7a. Scores will be tabulated from 0 to 35. A score of 35 represents a high level of pain medication misuse. A score of 0 represents a low level of pain medication misuse.
Post-operative Complication Rate | Post-operative days 0-90
  The researchers will review the electronic medical record to the rate and type of post-operative complications after ankle fracture surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Wilson, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis/Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
After deidentification, all individual participant data may be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning at the time of publication and ending 36 months after publication.
Access Criteria: Deidentified participant data will be shared with other investigators based on any reasonable request, as deemed appropriate by the study team. Requests may be submitted to Noah Harrison at nharrison@wustl.edu for review. Link to data will be provided at the time of request approval.

REFERENCES:
- [Background] Lawal OD, Gold J, Murthy A, Ruchi R, Bavry E, Hume AL, Lewkowitz AK, Brothers T, Wen X. Rate and Risk Factors Associated With Prolonged Opioid Use After Surgery: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Jun 1;3(6):e207367. doi: 10.1001/jamanetworkopen.2020.7367. PMID 32584407
- [Background] Vadivelu N, Hines RL. Buprenorphine: a unique opioid with broad clinical applications. J Opioid Manag. 2007 Jan-Feb;3(1):49-58. doi: 10.5055/jom.2007.0038. PMID 17367094
- [Background] Jasinski DR, Pevnick JS, Griffith JD. Human pharmacology and abuse potential of the analgesic buprenorphine: a potential agent for treating narcotic addiction. Arch Gen Psychiatry. 1978 Apr;35(4):501-16. doi: 10.1001/archpsyc.1978.01770280111012. PMID 215096
- [Background] Walsh SL, Babalonis S. The Abuse Potential of Prescription Opioids in Humans-Closing in on the First Century of Research. Curr Top Behav Neurosci. 2017;34:33-58. doi: 10.1007/7854_2016_448. PMID 27356522
- [Background] Walsh SL, Preston KL, Stitzer ML, Cone EJ, Bigelow GE. Clinical pharmacology of buprenorphine: ceiling effects at high doses. Clin Pharmacol Ther. 1994 May;55(5):569-80. doi: 10.1038/clpt.1994.71. PMID 8181201
- [Background] Kress HG. Clinical update on the pharmacology, efficacy and safety of transdermal buprenorphine. Eur J Pain. 2009 Mar;13(3):219-30. doi: 10.1016/j.ejpain.2008.04.011. Epub 2008 Jun 24. PMID 18567516
- [Background] Pergolizzi JV Jr, Magnusson P, LeQuang JA, Breve F, Mitchell K, Chopra M, Varrassi G. Transdermal Buprenorphine for Acute Pain in the Clinical Setting: A Narrative Review. J Pain Res. 2021 Mar 31;14:871-879. doi: 10.2147/JPR.S280572. eCollection 2021. PMID 33833565
- [Background] Desai SN, Badiger SV, Tokur SB, Naik PA. Safety and efficacy of transdermal buprenorphine versus oral tramadol for the treatment of post-operative pain following surgery for fracture neck of femur: A prospective, randomised clinical study. Indian J Anaesth. 2017 Mar;61(3):225-229. doi: 10.4103/ija.IJA_208_16. PMID 28405035
- [Background] Arshad Z, Prakash R, Gautam S, Kumar S. Comparison between Transdermal Buprenorphine and Transdermal Fentanyl for Postoperative Pain Relief after Major Abdominal Surgeries. J Clin Diagn Res. 2015 Dec;9(12):UC01-4. doi: 10.7860/JCDR/2015/16327.6917. Epub 2015 Dec 1. PMID 26816973
- [Background] Kim HJ, Ahn HS, Nam Y, Chang BS, Lee CK, Yeom JS. Comparative study of the efficacy of transdermal buprenorphine patches and prolonged-release tramadol tablets for postoperative pain control after spinal fusion surgery: a prospective, randomized controlled non-inferiority trial. Eur Spine J. 2017 Nov;26(11):2961-2968. doi: 10.1007/s00586-017-5213-5. Epub 2017 Jul 20. PMID 28730328
- [Background] Londhe S, Patwardhan M, Shah R, Oak M. Efficacy and Safety of Buprenorphine Transdermal Patch for Immediate Postoperative Analgesia After Total Knee Arthroplasty Surgery. J Arthroplasty. 2020 Jun;35(6S):S178-S181. doi: 10.1016/j.arth.2020.02.015. Epub 2020 Feb 13. PMID 32201109
- [Background] Londhe SB, Patwardhan M, Shah RV, Oak M, Shah A, Antao N, Khot R. Comparison of Efficacy and Safety of Transdermal Buprenorphine Patch and Conventional Analgesics in Intra-capsular Femur Neck Fracture Post Hemiarthroplasty. Indian J Orthop. 2022 Jun 25;56(8):1363-1369. doi: 10.1007/s43465-022-00668-7. eCollection 2022 Aug. PMID 35928664
- [Background] Niyogi S, Bhunia P, Nayak J, Santra S, Acharjee A, Chakraborty I. Efficacy of transdermal buprenorphine patch on post-operative pain relief after elective spinal instrumentation surgery. Indian J Anaesth. 2017 Nov;61(11):923-929. doi: 10.4103/ija.IJA_118_17. PMID 29217859
- [Background] Setti T, Sanfilippo F, Leykin Y. Transdermal buprenorphine for postoperative pain control in gynecological surgery: a prospective randomized study. Curr Med Res Opin. 2012 Oct;28(10):1597-608. doi: 10.1185/03007995.2012.719864. Epub 2012 Sep 10. PMID 22876835
- [Background] Xu X, Xie L, Liu H, Hu Y. Transdermal buprenorphine patch versus oral celecoxib for pain management after total knee arthroplasty: An open- label, randomized controlled trial. Orthop Traumatol Surg Res. 2020 Sep;106(5):915-919. doi: 10.1016/j.otsr.2020.04.010. Epub 2020 Jul 2. PMID 32624377
- [Background] Burden M, Keniston A, Wallace MA, Busse JW, Casademont J, Chadaga SR, Chandrasekaran S, Cicardi M, Cunningham JM, Filella D, Hoody D, Hilden D, Hsieh MJ, Lee YS, Melley DD, Munoa A, Perego F, Shu CC, Sohn CH, Spence J, Thurman L, Towns CR, You J, Zocchi L, Albert RK. Opioid Utilization and Perception of Pain Control in Hospitalized Patients: A Cross-Sectional Study of 11 Sites in 8 Countries. J Hosp Med. 2019 Dec 1;14(12):737-745. doi: 10.12788/jhm.3256. Epub 2019 Jul 24. PMID 31339840
- [Background] Otwell AG, Stambough JB, Cherney SM, Blake L, Siegel ER, Mears SC. Does the type of lower extremity fracture affect long-term opioid usage? A meta-analysis. Arch Orthop Trauma Surg. 2024 Mar;144(3):1221-1231. doi: 10.1007/s00402-023-05174-5. Epub 2024 Feb 16. PMID 38366036
- [Background] Skibicki H, Saini S, Rogero R, Nicholson K, Shakked RJ, Fuchs D, Winters BS, Raikin SM, Pedowitz DI, Daniel JN. Opioid Consumption Patterns and Prolonged Opioid Use Among Opioid-Naive Ankle Fracture Patients. Foot Ankle Spec. 2023 Feb;16(1):36-42. doi: 10.1177/1938640021992922. Epub 2021 Feb 12. PMID 33576251
- [Background] Yokell MA, Zaller ND, Green TC, Rich JD. Buprenorphine and buprenorphine/naloxone diversion, misuse, and illicit use: an international review. Curr Drug Abuse Rev. 2011 Mar;4(1):28-41. doi: 10.2174/1874473711104010028. PMID 21466501
- [Background] Carl P, Crawford ME, Madsen NB, Ravlo O, Bach V, Larsen AI. Pain relief after major abdominal surgery: a double-blind controlled comparison of sublingual buprenorphine, intramuscular buprenorphine, and intramuscular meperidine. Anesth Analg. 1987 Feb;66(2):142-6. PMID 3544957
- [Background] Dobkin AB, Esposito B, Philbin C. Double-blind evaluation of buprenorphine hydrochloride for post-operative pain. Can Anaesth Soc J. 1977 Mar;24(2):195-202. doi: 10.1007/BF03006232. PMID 321103
- [Background] Chakravarty K, Tucker W, Rosen M, Vickers MD. Comparison of buprenorphine and pethidine given intravenously on demand to relieve postoperative pain. Br Med J. 1979 Oct 13;2(6195):895-7. doi: 10.1136/bmj.2.6195.895. PMID 391321
- [Background] Tigerstedt I, Tammisto T. Double-blind, multiple-dose comparison of buprenorphine and morphine in postoperative pain. Acta Anaesthesiol Scand. 1980 Dec;24(6):462-8. doi: 10.1111/j.1399-6576.1980.tb01584.x. PMID 7018155
- [Background] Masson AH. Sublingual buprenorphine versus oral dihydrocodeine in post-operative pain. J Int Med Res. 1981;9(6):506-10. doi: 10.1177/030006058100900614. PMID 7319134
- [Background] Mok MS, Lippmann M, Steen SN. Multidose/observational, comparative clinical analgetic evaluation of buprenorphine. J Clin Pharmacol. 1981 Jul;21(7):323-9. doi: 10.1002/j.1552-4604.1981.tb01774.x. PMID 7263931
- [Background] Ouellette RD. Buprenorphine and morphine efficacy in postoperative pain: a double-blind multiple-dose study. J Clin Pharmacol. 1982 Apr;22(4):165-72. doi: 10.1002/j.1552-4604.1982.tb02158.x. PMID 7047580
- [Background] Freedman M. A comparison of buprenorphine and pentazocine for the relief of postoperative pain. S Afr Med J. 1986 Jan 4;69(1):27-8. PMID 3510458
- [Background] Maunuksela EL, Korpela R, Olkkola KT. Comparison of buprenorphine with morphine in the treatment of postoperative pain in children. Anesth Analg. 1988 Mar;67(3):233-9. PMID 3344976
- [Background] Maunuksela EL, Korpela R, Olkkola KT. Double-blind, multiple-dose comparison of buprenorphine and morphine in postoperative pain of children. Br J Anaesth. 1988 Jan;60(1):48-55. doi: 10.1093/bja/60.1.48. PMID 3337794
- [Background] Dingus DJ, Sherman JC, Rogers DA, DiPiro JT, May R, Bowden TA Jr. Buprenorphine versus morphine for patient-controlled analgesia after cholecystectomy. Surg Gynecol Obstet. 1993 Jul;177(1):1-6. PMID 8322143
- [Background] Khandelwal H, Negi A, Govil N, Singh A, Parag K, Bhardwaj BB. Comparative evaluation of analgesic efficacy of buprenorphine transdermal patch and fentanyl patch in management of postoperative pain after arthroscopic lower limb surgery: A randomized controlled trial. J Anaesthesiol Clin Pharmacol. 2021 Apr-Jun;37(2):272-278. doi: 10.4103/joacp.JOACP_405_20. Epub 2021 Jul 15. PMID 34349379
- [Background] Lee JH, Kim JH, Kim JH, Kim HS, Min WK, Park YS, Lee KY, Lee JH. Efficacy and Safety of Transdermal Buprenorphine versus Oral Tramadol/Acetaminophen in Patients with Persistent Postoperative Pain after Spinal Surgery. Pain Res Manag. 2017;2017:2071494. doi: 10.1155/2017/2071494. Epub 2017 Sep 13. PMID 29056859